CLINICAL TRIAL: NCT03780842
Title: Effect of Changing Levels of Neurally Adjusted Ventilatory Assist (NAVA) on Respiratory Parameters in Newborns Receiving NAVA Ventilation
Brief Title: Effect of Changing Levels of Neurally Adjusted Ventilatory Assist (NAVA) in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Lefevere (Other)
Responsible Party: Sponsor-Investigator, Julie Lefevere, Resident, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pilot breakpoint NAVA
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Newborn Morbidity

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, exploratory study in a convenience sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invasive NAVA ventilation (Experimental): A titration protocol will be used for changing NAVA levels in intubated newborns
  Interventions: Device: NAVA level
- Non-invasive NAVA ventilation (Experimental): A titration protocol will be used for changing NAVA levels in newborns with non-invasive NAVA ventilation (= with a nasal interface).
  Interventions: Device: NAVA level

INTERVENTIONS:
Device: NAVA level — A titration protocol will be used for changing NAVA levels. The NAVA level will be reduced to 0,5 cmH2O/µV for 3 minutes as a starting point. Limit peak pressure will be set to 35cmH2O (i.e. according to the standard manufacturer's settings) the maximum pressure that can be delivered to the patient is cut off at 30cmH2O). Other ventilator settings will be left unchanged and are as clinically indicated. Ventilator settings will be according to our standard of care and as following: PEEP between 4 and 7 mmHg, apnea time 2-5 sec, back-up ventilation with a pressure above PEEP between 5 and 15 mmHg and a frequency between 30 and 50 per minute.
  Starting from a NAVA level of 0,5 cmH20/µV the level will be increased by 0,5 cmH2O/µV every 3 minutes until reaching a maximum NAVA level of 4,0 cmH2O/µV.

SUMMARY:
To examine the effect of changing levels of support during NAVA-ventilation ("NAVA-level") on electrical diaphragm activity of the newborn on invasive or non-invasive NAVA ventilation.

The aim is to explore whether a so-called 'breakpoint', as defined in previous studies on NAVA ventilation in adults and children(1, 9), can be determined in newborn infants. Knowledge of this breakpoint will be used to optimise the settings of NAVA level at initiation of invasive or non-invasive NAVA ventilation.

This is an explorative study conducted in preparation of a randomized controlled trial that is planned in the near future to compare the effects of non-invasive NAVA with nasal continuous positive airway pressure (CPAP) in newborn infants.

ELIGIBILITY:
Inclusion Criteria:

* Newborns admitted to the NICU in need for respiratory support and put on invasive or non-invasive NAVA by the attending physician. Patients will be included when they are clinically stable and within 24h after starting NAVA or nivNAVA.

Exclusion Criteria:

* - Congenital malformations of the diaphragm or respiratory system, including congenital diaphragmatic hernia.
* Patients with abnormalities of the upper airway (e.g. vocal cord paralysis, post-extubation laryngeal edema, Pierre-Robin sequence…).
* More than 20% of time spent in back-up ventilationWhen a patient on NAVA ventilation is apneic for a certain period of time (apnea time), the ventilator switches tot backup-ventilation. Backup-ventilation is pressure controlled, the apnea time can variate between 2 and 10 seconds.
* Clinically unstable patients:
* hemodynamic instability as defined by need of inotropic support or
* rapid respiratory deterioration on NAVA ventilation.
* No informed consent.

Max Age: 20 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Optimal NAVA level to unload the diaphragm | 24 minutes
  The aim is to explore whether a so-called 'breakpoint', as defined in previous studies on NAVA ventilation in adults and children(1, 9), can be determined in newborn infants. Knowledge of this breakpoint will be used to optimise the settings of NAVA level at initiation of invasive or non-invasive NAVA ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lefevere J, Van Delft B, Vervoort M, Cools W, Cools F. Non-invasive neurally adjusted ventilatory assist in preterm infants with RDS: effect of changing NAVA levels. Eur J Pediatr. 2022 Feb;181(2):701-707. doi: 10.1007/s00431-021-04244-3. Epub 2021 Sep 17. PMID 34533644